CLINICAL TRIAL: NCT03098238
Title: Endothelial Microparticules as Biomarker of Antibody-mediated Rejection in Kidney Transplantation
Brief Title: Endothelial Microparticules and Antibody Mediated Rejection and Kidney Transplantation: Biomarker of Antibody-mediated Rejection in Kidney Transplantation
Acronym: MICROMARK RJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RECHMPL16_0263; UF 9746 (Other: Montpellier University Hospital)
Record Dates: First submitted 2017-03-26; First posted 2017-03-31 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2020-01

CONDITIONS: Renal Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients without humoral rejection or DSA (Other): Renal transplant patients with systematic kidney biopsy at 3 months and 12 months Patients without humoral rejection or DSA (Donor Specific Antibodies)
  Interventions: Biological: Biological sample
- Patient without humoral rejection with a DSA (Other): Patient without humoral rejection with a DSA (Donor Specific Antibodies)Patients with a graft biopsy for a donor-specific anti-HLA antibody
  Interventions: Biological: Biological sample
- Patients with humoral rejection (Other): Patients with humoral rejection
  Interventions: Biological: Biological sample

INTERVENTIONS:
Biological: Biological sample — Biological sampling of two citrate tubes (18 ml) during a normal blood

SUMMARY:
Context and rationale:

Antibody-mediated rejection is the leading cause of long-term renal graft loss. It's due to the production by the recipient of antibodies directed against antigens (belonging or not to the HLA system) present on the surface of the donor specific endothelial cells (DSA), leading to graft failure.

The main difficulty to manage the humoral rejection is the delay of the diagnosis and the treatment to slow the evolution towards fibrosis.

Positivity of anti-HLA antibodies is the main risk factor for the rejection but the only way to make the diagnosis of humoral rejection is to perform a graft biopsy, an invasive process.

Endothelial microparticles (MPE) are small membrane vesicles generated by endothelial cell activation and / or apoptosis processes.

We test the hypothesis that endothelial microparticles are an early diagnostic biomarker of humoral rejection in renal transplantation allowing to detect it at the "subclinical" stage.

Primary and secondary objectives:

The main objective of this study is to estimate the performance of MPE plasma concentration for the diagnosis of humoral rejection in renal transplant patients with DSA. The secondary objective is to investigate by mass spectrometry the MPEs specific to the endothelium of the graft and to evaluate their diagnostic performance in relation to non-specific MEPs

Methodology :

We will conduct a cross-sectional evaluation of a diagnostic method from a collection of biological samples. The gold standard for the diagnosis of humoral rejection is the histological diagnosis on graft biopsy. The new test under study will be the flow cytometric assay of the MPE concentration carried out on plasma taken on the day of the graft biopsy.

Feasibility:

Among the active list of renal transplant patients attending the Montpellier University Hospital, we estimate that we can include the number of subjects required (N = 250) over 18 months. This work will be carried out in a laboratory with all the tools and techniques used, in particular flow cytometry and mass spectrometry, perfectly mastered and realized on dedicated technical platforms

Benefits / Outlook:

find a non-invasive early diagnostic biomarker to detect humoral rejection from the "subclinical" stage in order to set up an adapted treatment as quickly as possible.

DETAILED DESCRIPTION:
Context and rationale:

Antibody-mediated rejection is the leading cause of long-term renal graft loss. It's due to the production by the recipient of antibodies directed against antigens (belonging or not to the HLA system) present on the surface of the donor specific endothelial cells (DSA), the binding of which can activate the renal endothelium and be responsible for inflammation leading to fibrosis and graft destruction.

The main obstacle in the management of the humoral rejection is the delay of the diagnosis and the treatment to slow the evolution towards fibrosis. At the beginning of the process there is no "apparent" dysfunction of the graft (elevation of serum creatinine and / or proteinuria) but only inflammation of the renal parenchyma: this is referred to as "subclinical" humoral rejection. Graft dysfunction occurs only when the inflammation is serious and responsible for irreversible lesions of fibrosis.

New sensitive detection techniques for anti-HLA antibodies allow to detect DSA well before the onset of humoral rejection but the only way to make the diagnosis of humoral rejection is to perform a graft biopsy, an invasive process with a hemorrhagic risk which can not be repeated too frequently.

Endothelial microparticles (MPE) are small membrane vesicles generated by endothelial cell activation and / or apoptosis processes. An increasing level in circulating blood appears today as a endothelial dysfunction in many pathologies. Their role in humoral rejection, a model of endothelial dysfunction, has never been explored.

We wish to test the hypothesis that endothelial microparticles are an early diagnostic biomarker of humoral rejection in renal transplantation allowing to detect it at the "subclinical" stage.

Primary and secondary objectives:

The main objective of this study is to estimate the performance of MPE plasma concentration for the diagnosis of humoral rejection in renal transplant patients with DSA. The secondary objective is to investigate by mass spectrometry the MPEs specific to the endothelium of the graft and to evaluate their diagnostic performance in relation to non-specific MEPs

Methodology :

We will conduct a cross-sectional evaluation of a diagnostic method from a collection of biological samples. The gold standard for the diagnosis of humoral rejection is the histological diagnosis on graft biopsy. The new test under study will be the flow cytometric assay of the MPE concentration carried out on plasma taken on the day of the graft biopsy.

Feasibility:

Among the active list of renal transplant patients attending the Montpellier University Hospital, we estimate that we can include the number of subjects required (N = 250) over 18 months. This work will be carried out in a laboratory with all the tools and techniques used, in particular flow cytometry and mass spectrometry, perfectly mastered and realized on dedicated technical platforms

Benefits / Outlook:

At a time when the shortage of organs is growing and becomes a real public health problem, it becomes essential to better control the management of humoral rejection, the main cause of long-term renal graft loss. One of the key steps in this step is to find a non-invasive early diagnostic biomarker to detect humoral rejection from the "subclinical" stage in order to set up an adapted treatment as quickly as possible.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at time of inclusion
* Renal transplant patients monitored at Montpellier University Hospital
* With a recent or planned realization of a graft biopsy
* Patients with DSA (s) detected by Single Antigen Bead Assay (SAB, LabScreen Single Antigen, One Lambda Kit) with an average fluorescence intensity> 500 IU Or Patients without DSA transplanted to a year with a systematic biopsy aspiration.

Exclusion Criteria:

* Refusal to participate in or to undergo the examination
* Major protected by guardianship
* History of treated humoral rejection
* Incompatible graft ABO
* Multi-organ transplantation
* Cardiovascular disease active (myocardial infarction <3 months, arteriopathy obliterating lower limbs stage III or IV)
* Sepsis in progress
* Evolving Cancers
* Lupus nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of endothelial microparticles | 1 day
  Endothelial microparticle (MPE) plasma concentration for the diagnosis of humoral rejection in renal transplant patients with DSA.

SECONDARY OUTCOMES:
Presence of specific MEPs | 1 day
  Presence of MPEs specific to the graft endothelium and to evaluate their diagnostic performance in relation to non-specific MEPs

CONTACTS AND LOCATIONS:
Overall Officials: Moglie LE QUINTREC DONNETTE, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC